CLINICAL TRIAL: NCT04884321
Title: Adults' Attitudes Toward Complementary And Alternative Medicine And Their State Of Using Complementary And Alternative Medicine During The COVID-19 Pandemic
Brief Title: Complementary And Alternative Medicine During The COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: Filiz Polat (Unknown); Aynur Ekren Çakıcı (Unknown)
Responsible Party: Principal Investigator, Leyla Delibas, Assistant Professor, Hasan Kalyoncu University
Other Study IDs: HasanKUMYO
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Complementary Therapies
Keywords: Complementary Therapies; COVID-19; Complementary and Alternative Medicine; Attitude
MeSH Terms: conditions — COVID-19; Behavior | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Complementary And Alternative Medicine — No intervention was done in the cross-sectional study

SUMMARY:
Complementary and alternative medicine is frequently used in the treatment of several groups of diseases.

DETAILED DESCRIPTION:
This study aimed to explore the attitudes of adults living in Turkey toward complementary and alternative medicine in the period of the COVID-19 pandemic and identify whether Turkish adults used it during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* agree to participate in the study
* not to be a communication problem

Exclusion Criteria:

* be a communication problem

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The research population was comprised of Turkish citizens who resided in Turkey and were aged 18-65 years.
Sampling Method: Non-Probability Sample
Enrollment: 3242 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Participant adults' responses to the questions raised about the use of complementary and alternative methods during the COVID-19 pandemic | 2021
Means of scores obtained by participant adults from the holistic complementary and alternative medicine questionnaire (HCAMQ) and its sub-scales | 2021
  Holistic Complementary and Alternative Medicine Questionnaire
Complementary and alternative treatment methods used during the COVID-19 pandemic | 2021
Plants consumed during the COVID-19 pandemic | 2021
Symptoms against which complementary and alternative methods are used during the COVID-19 pandemic | 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Ünivrsitesi, Gaziantep, Lütfen Seç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided